CLINICAL TRIAL: NCT00758862
Title: The Pharmacokinetics of 2% TD1414 Cream in Adults With Secondarily Infected Traumatic Lesions (SITL) or Impetigo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TD1414-C22
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2018-06

CONDITIONS: Secondarily Infected Traumatic Lesions (SITL); Impetigo
MeSH Terms: conditions — Impetigo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: 2% TD1414 Cream

INTERVENTIONS:
Drug: 2% TD1414 Cream — Application 3 times daily for 7 days

SUMMARY:
A national, prospective single arm phase II study investigating the pharmacokinetics and safety of the 2% TD1414 cream when applied 3 times daily for 7 days to adult patients with impetigo or Secondarily Infected Traumatic Lesions (SITL). A total of 20 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to comply with all the study requirements/procedures
* Age ≥ 18 and ≤65 years
* Primary bullous/non-bullous impetigo or SITL
* Patients suffering from primary bullous/non-bullous impetigo must have:

  * Not more than 10 discrete lesions, and
  * A total lesional area ≥ 1 cm2 and ≤ 100 cm2, and
  * Any surrounding erythema must not extend beyond 2 cm from the edge of the lesion, and
  * Total SIRS score equal to or ≥ 8
* Patients suffering from SITL must have:

  * A total infected area of the traumatic lesion ≥ 1 cm2 and ≤ 100 cm2, and
  * Any surrounding erythema must not extend beyond 2 cm from the edge of the lesion, and
  * Total SIRS score ≥ 8, and
  * SITL not caused by burns or animal/human bite
* Amenable for treatment with topical antibiotic alone
* Body Mass Index ≥18 and ≤ 35 kg/m2.

Exclusion Criteria:

* Immunosuppressed state or other serious systemic disease
* Signs and/or symptoms of systemic infection, such as malaise and fever or local adenopathy and fever
* Unwillingness to abstain from use of any other topical products including emollients on the lesional area during the study
* Systemic treatment with antibacterials or immunosuppressive agents (e.g. corticosteroids) within 2 days before day 1 (inhaled/intranasal steroids may be used)
* Topical treatment with antibacterials, immunosuppressive agents (e.g. corticosteroids) or antiseptics (e.g. alcohol, chlorhexidine, hydrogen peroxide, iodine) on the lesional area within 2 days before day 1
* Indication for surgical or systemic treatment of the SITL/impetigo
* Known or suspected hypersensitivity to any of the components of the study medication
* Participation in any other interventional clinical trial or use of an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to day 1
* Previously enrolled in this study
* A blood alcohol content ≥ 0.08% as determined by a Breathalyzer test
* Known or suspected history of alcohol abuse/alcoholism or drug abuse
* Known or suspected impairment of liver function
* Heart rhythm disturbances or clinically significant quantitative or qualitative abnormality in the pretreatment ECG
* Blood donation in excess of 500mL within 56 days before day 1 or donation during the study or within 3 days of leaving the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terry Jones, MD, Principal Investigator — J&S Studies Inc.
Locations (1):
- J&S Studies, Inc., College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- TD1414: 2% TD1414 Cream: Application 3 times on lesions area(s) daily for 7 days. A maximum of 0.5g of cream on a 100 cm2 lesion area was to be used per application.
Period: Overall Study
Arm/Group | TD1414
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- TD1414: 2% TD1414 Cream: Application 3 times daily for 7 days
Arm/Group | TD1414
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: TD1414 Serum Concentration by Timepoint
Description: On Days 1 and 2(and possibly Day 3 depending on the time of first application on Day 1) a sample was taken for pharmacokinetic(PK) analysis at any time before first application on Day 1, and at 12±1, 18±1, 24±1 and 36±4 hours after first application. If the 36±4 hours sampling time fell on Day 3, then a second sample was also required on Day 3, but was to be obtained at 6pm or afterwards. On Days 3 to 6(and also Day 7 if the very last application fell on Day 8), one sample was taken on each day at any time during the day. On Days 7 and 8(or Days 8 and 9 if very last application was on Day 8), a sample was taken immediately before the very last application and at 6±1, 12±1 and 24±2 hours after the very last application. On Days 9 and 10, one sample was taken on each day at any time during the day. If the participant had already had a sample(s) taken on Day 9 because the timing of some of the post-last application samples fell on this day, then further samples were not required on Day 9
Time Frame: From 0 hours to 240 hours
Population: One participant withdrew at day 3 due to the participant being out of range of the inclusion criterion.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | TD1414
Number analyzed (Participants) | 20
pg/mL
  12 hours Post First Application | 624.3 (1255.3)
  18 hours Post First Application | 864.1 (1635.7)
  24 hours Post First Application | 1195.7 (2448.1)
  36 hours Post First Application | 888.4 (1878.6)
  Day 3 | 659.1 (1461.8)
  Day 4: number analyzed (Participants) | 19
  Day 4 | 309.0 (578.5)
  Day 5: number analyzed (Participants) | 19
  Day 5 | 344.4 (673.0)
  Day 6: number analyzed (Participants) | 19
  Day 6 | 178.8 (199.1)
  Prior last application: number analyzed (Participants) | 19
  Prior last application | 177.4 (220.5)
  6 hours Post Last Application: number analyzed (Participants) | 19
  6 hours Post Last Application | 189.9 (231.1)
  12 hours Post Last Application: number analyzed (Participants) | 19
  12 hours Post Last Application | 190.6 (214.0)
  24 hours Post Last Application: number analyzed (Participants) | 19
  24 hours Post Last Application | 108.6 (135.0)
  Day 9: number analyzed (Participants) | 19
  Day 9 | 99.2 (125.4)
  Day 10: number analyzed (Participants) | 19
  Day 10 | 47.2 (60.1)

2. Primary Outcome: Peak TD1414 Serum Concentration (Cmax )
Description: The Cmax was summarised by lesion size at baseline, by SIRS scores at baseline and by amount of TD1414 cream used.
  Please see 1. Primary Outcome for details on collection of blood samples for the Pharmacokinetic analyses. For description of lesion size, SIRS score and amount of TD1414 cream used please see outcome measure 3, 4 and 5 respectively.
Time Frame: From 0 hours to 240 hours
Population: Cmax could not be calculated for one participant as all values below lower limit of quantification (TD1414 concentration = 50pg/mL).
Measure: Geometric Mean (Standard Deviation); unit: pg/mL
Arm/Group | TD1414
Number analyzed (Participants) | 20
pg/mL | 650.4 (2433.6)

3. Primary Outcome: Peak Serum Concentration by Baseline Lesion Size
Description: On Day 1 (before the first application), the (sub)investigator recorded the size of the lesion(s). For each participant the size of the lesion was allocated to one of two categories: ≤15cm² or >15cm². The Cmax is presented by baseline lesion size category (≤15 cm² and >15 cm²).
  Please see 1. Primary Outcome for details on collection of blood samples for the Pharmacokinetic analyses.
Time Frame: From 0 hours to 240 hours
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: pg/mL
Arm/Group | TD1414
Number analyzed (Participants) | 20
pg/mL
  <=15 cm^2: number analyzed (Participants) | 13
  <=15 cm^2 | 484.1 (1755.1)
  >15 cm^2: number analyzed (Participants) | 6
  >15 cm^2 | 1233.3 (3545.0)

4. Primary Outcome: Peak Serum Concentration by SIRS Score
Description: On Day 1 (before the first application), the (sub)investigator recorded the severity of the lesion(s).
  The severity was to be recorded using the Severity of Infection Rating Scale (SIRS).
  For the SIRS, the following seven clinical signs/symptoms of infection were assessed:
  Exudates/pus Crusting Erythema Oedema Tissue warmth Itching Pain
  Each of the seven signs/symptoms was scored using the following scale:
  0 = absent 2 = mild 4 = moderate 6 = severe The scores for each sign/symptom were summed to give the total SIRS score. The total SIRS score could range from 0 to 42.
  Please see 1. Primary Outcome for details on collection of blood samples for the Pharmacokinetic analyses.
Time Frame: From 0 hours to 240 hours
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: pg/mL
Arm/Group | TD1414
Number analyzed (Participants) | 20
pg/mL
  SIRS score <=13: number analyzed (Participants) | 10
  SIRS score <=13 | 416.2 (1937.5)
  SIRS score >13: number analyzed (Participants) | 9
  SIRS score >13 | 1068.3 (2931.6)

5. Primary Outcome: Peak Serum Concentration by Amount of TD1414 Cream Used
Description: The weight of TD1414 cream used was calculated by subtracting the weight of the used dispensed tube from the mean weight of a full tube.
  Please see 1. Primary Outcome for details on collection of blood samples for the Pharmacokinetic analyses.
Time Frame: From 0 hours to 240 hours
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: pg/mL
Arm/Group | TD1414
Number analyzed (Participants) | 20
pg/mL
  <=2 g: number analyzed (Participants) | 8
  <=2 g | 323.5 (858.2)
  >2 g: number analyzed (Participants) | 11
  >2 g | 1081.0 (2976.6)

6. Primary Outcome: Time to Reach Peak Serum Concentration (Tmax )
Description: Please see 1. Primary Outcome for details on collection of blood samples for the Pharmacokinetic analyses.
Time Frame: From 0 hours to 240 hours
Population: Tmax could not be calculated for one participant as all values below lower limit of quantification (TD1414 concentration = 50pg/mL).
Measure: Median (Standard Deviation); unit: hours
Arm/Group | TD1414
Number analyzed (Participants) | 20
hours | 32.08 (59.82)

7. Primary Outcome: Time to Reach Peak Serum Concentration (Tmax ) by Baseline Lesion Size
Description: Please see 1. Primary Outcome for details on collection of blood samples for the Pharmacokinetic analyses.
Time Frame: From 0 hours to 240 hours
Population: as for outcome 6
Measure: Median (Standard Deviation); unit: hours
Arm/Group | TD1414
Number analyzed (Participants) | 20
hours
  <=15 cm^2: number analyzed (Participants) | 13
  <=15 cm^2 | 47.42 (56.91)
  >15 cm^2: number analyzed (Participants) | 6
  >15 cm^2 | 23.73 (69.77)

8. Primary Outcome: Time to Reach Peak Serum Concentration (Tmax ) by SIRS Score
Description: Please see 1. Primary Outcome for details on collection of blood samples for the Pharmacokinetic analyses.
Time Frame: From 0 hours to 240 hours
Population: AUC(0-t) could not be calculated for one participant as all values below lower limit of quantification (TD1414 concentration = 50pg/mL).
Measure: Median (Standard Deviation); unit: hours
Arm/Group | TD1414
Number analyzed (Participants) | 20
hours
  <=13 cm^2: number analyzed (Participants) | 10
  <=13 cm^2 | 42.21 (62.79)
  >13 cm^2: number analyzed (Participants) | 9
  >13 cm^2 | 24.22 (58.03)

9. Primary Outcome: Time to Reach Peak Serum Concentration (Tmax ) by Amount of TD1414 Cream Used
Description: Please see 1. Primary Outcome for details on collection of blood samples for the Pharmacokinetic analyses.
Time Frame: From 0 hours to 240 hours
Population: as for outcome 6
Measure: Median (Standard Deviation); unit: hours
Arm/Group | TD1414
Number analyzed (Participants) | 20
hours
  <=2 g: number analyzed (Participants) | 8
  <=2 g | 28.15 (63.90)
  >2 g: number analyzed (Participants) | 11
  >2 g | 33.65 (62.68)

10. Primary Outcome: Area Under the Curve (AUC(0-t))
Description: Area under the concentration-time curve (AUC(0-t)) from time 0 to time of last non-zero observation after dosing, calculated by linear/log trapezoidal method.
  Please see 1. Primary Outcome for details on collection of blood samples for the Pharmacokinetic analyses.
Time Frame: From 0 hours to 240 hours
Population: as for outcome 8
Measure: Geometric Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | TD1414
Number analyzed (Participants) | 20
h*pg/mL | 32138 (123032)

11. Primary Outcome: Area Under the Curve by Baseline Lesion Size
Description: On Day 1 (before the first application), the (sub)investigator recorded the size of the lesion(s). For each participant the size of the lesion was allocated to one of two categories: ≤15cm² or >15cm².
  Please see 1. Primary Outcome for details on collection of blood samples for the Pharmacokinetic analyses.
Time Frame: From 0 hours to 240 hours
Population: as for outcome 8
Measure: Geometric Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | TD1414
Number analyzed (Participants) | 20
h*pg/mL
  <=15 cm^2: number analyzed (Participants) | 13
  <=15 cm^2 | 21240 (61954)
  >15 cm^2: number analyzed (Participants) | 6
  >15 cm^2 | 78836 (192236)

12. Primary Outcome: Area Under the Curve by SIRS Score
Description: On Day 1 (before the first application), the (sub)investigator recorded the severity of the lesion(s).
  The severity was to be recorded using the Severity of Infection Rating Scale (SIRS).
  For the SIRS, the following seven clinical signs/symptoms of infection were assessed:
  Exudates/pus, Crusting, Erythema, Oedema, Tissue warmth, Itching and Pain.
  Each of the seven signs/symptoms was scored using the following scale:
  0 = absent 2 = mild 4 = moderate 6 = severe
  The scores for each sign/symptom were summed to give the total SIRS score. The total SIRS score could range from 0 to 42.
  Please see 1. Primary Outcome for details on collection of blood samples for the Pharmacokinetic analyses.
Time Frame: From 0 hours to 240 hours
Population: as for outcome 8
Measure: Geometric Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | TD1414
Number analyzed (Participants) | 20
h*pg/mL
  SIRS score <=13: number analyzed (Participants) | 10
  SIRS score <=13 | 17923 (69972)
  SIRS score >13: number analyzed (Participants) | 9
  SIRS score >13 | 61488 (160681)

13. Primary Outcome: Area Under the Curve (AUC(0-t)) by Amount of TD1414 Cream Used
Description: as for outcome 5
Time Frame: From 0 hours to 240 hours
Population: as for outcome 8
Measure: Geometric Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | TD1414
Number analyzed (Participants) | 20
h*pg/mL
  <=2 g: number analyzed (Participants) | 8
  <=2 g | 13642 (23828)
  >2 g: number analyzed (Participants) | 11
  >2 g | 59932 (150278)

ADVERSE EVENTS:
Time Frame: From Day 1 to Day 10
Arm/Group | TD1414
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Company acknowledges the investigator's right to publish the entire results of the study, irrespective of outcome. The Company retains the right to have any publication submitted to the Company for review at least 30 days prior to the same paper being submitted for publication or presentation. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.